CLINICAL TRIAL: NCT01738932
Title: Genetic Polymorphisms of Mannan-binding Lectin (MBL) and Serum Levels of MBL in Patients With Endometriosis
Brief Title: Genetic Polymorphisms of Mannan-binding Lectin (MBL)and Serum Levels of MBL in Patients With Endometriosis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MBLendo06
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Endometriosis
Keywords: endometriosis; mannan-binding lectin; immunology
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, EDTA blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: women with histologically verified endometriosis
- Controls: Healthy Danish blood donors

SUMMARY:
The purpose of the study is to investigate the possible association between low levels of MBL and the development of endometriosis

DETAILED DESCRIPTION:
Endometriosis is a chronic, inflammatory disease, affecting approximately 10% of the female population. The pathogenesis of endometriosis is still unclear, but several studies have indicated that the immune system is involved. It has been suggested that endometriosis should be considered an autoimmune disease, considering the findings of elevated levels of cytokines, decreased cell apoptosis, increased incidence of autoantibodies and a higher frequency of other autoimmune diseases in endometriosis patients. MBL participates in the innate immune defence by activating complement on the surfaces of microorganisms, but several studies have suggested that MBL is also involved in autoimmune diseases. The individual MBL level is highly variable due to a number of polymorphic sites in the structural gene and in the promoter region, and approximately 12 % of the normal population have very low serum MBL levels (<100 ng/ml).

The possible association between MBL and endometriosis has been investigated in two small studies, in which no association was found. The aim of the present study is to investigate the prevalence of individuals with low serum levels of MBL and with genotypes associated with low MBL production in a larger group of endometriosis patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified endometriosis
* ASRM stage 2-4

Exclusion Criteria:

* pregnancy
* actual treatment with GnRh analog
* autoimmune diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Endometriosis patients referred to the endometriosis clinic at Aarhus University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Frequency of individuals with s-MBL < 100 ng/ml | baseline
Frequency of individuals with MBL genotypes LXPA/O or O/O | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kruse, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Gynecology and Obstetrics, Aarhus, Denmark

REFERENCES:
- [Result] Kavoussi SK, Mueller MD, Lebovic DI. Expression of mannose-binding lectin in the peritoneal fluid of women with and without endometriosis. Fertil Steril. 2006 May;85(5):1526-8. doi: 10.1016/j.fertnstert.2005.10.032. Epub 2006 Apr 5. PMID 16600231
- [Result] Ozerkan K, Oral B, Uncu G. Mannose-binding lectin levels in endometriosis. Fertil Steril. 2010 Jul;94(2):775-6. doi: 10.1016/j.fertnstert.2009.09.056. Epub 2009 Nov 14. PMID 19917506